CLINICAL TRIAL: NCT00540202
Title: Effectiveness of Oral Quinine and Artemether-Lumefantrine in the Treatment of Uncomplicated Malaria in Ugandan Children
Acronym: QALE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Ministry of Health, Uganda (Other Government); Uganda Malaria Surveillance Project (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QALE07
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Uncomplicated Malaria
Keywords: Effectiveness; Oral quinine; Coartem; Uncomplicated malaria; Children
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.Oral quinine (Experimental): Patients will be given oral quinine at the dose of 10mg/kg 8 hourly for 7 days
  Interventions: Drug: Oral quinine
- 2. Coartem (Active Comparator): Tablets
  Interventions: Drug: artemether-lumefantrine

INTERVENTIONS:
Drug: artemether-lumefantrine — Tablets taken twice daily for 3 days according to weight based guidelines.
  Other Names: Coartem
  Arms: 2. Coartem
Drug: Oral quinine — Quinine tablets given at 10mg/kg 8 hourly for 7 days
  Arms: 1.Oral quinine

SUMMARY:
We will test the hypothesis that there is a difference in effectiveness of oral quinine in comparison to artemether Lumefantrine in the treatment of uncomplicated malaria in children.

DETAILED DESCRIPTION:
This study will be designed as an open randomized effectiveness study assessing the parasitological and clinical cure rates and adherence to oral quinine monotherapy in comparison to artemether-Lumefantrine. We will also describe some of the adverse events to the two drugs.The measurements will include age, sex, weight, hemoglobin levels on days 0, 7, 14 and 28, parasite density on days 0, 7, 14 and 28 and clinical examination findings. Adverse events will also be documented

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 6 and 59 months of age seen at the assessment centre during the study period
2. With fever defined as axillary temperature ≥37.5 °C or history of fever in the past 24 h
3. With a microscopically confirmed monoinfection of Plasmodium falciparum
4. Able to tolerate oral therapy,
5. Whose parents/guardians have provided written informed consent.

Exclusion Criteria:

1. Children with a history of allergy to quinine, artemether-Lumefantrine or milk.
2. Evidence of severe malaria.
3. Residence at more than 20km from the health clinic.
4. Evidence of a significant concomitant febrile illness that would require hospitalization or chronic medical illness

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Estimated)
Dates: Start 2007-09; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
1. PCR adjusted parasitological cure rate on day 28. 2. Clinical cure rates on day 28. | 28 days

SECONDARY OUTCOMES:
1. Fever clearance time assessed by self report. 2. Hemoglobin changes on day 0, 7, 14 and 28. 3. Safety profiles. 4. Adherence: measured by patient report and pill count on day 3 for the artemether-Lumefantrine group and day 7 for the quinine group. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose O Talisuna, PhD, Principal Investigator — Ministry of Health, Uganda
Locations (1):
- Mulago National Referral Hospital, Kampala, Central Region, Uganda

REFERENCES:
- [Background] Fogg C, Bajunirwe F, Piola P, Biraro S, Checchi F, Kiguli J, Namiiro P, Musabe J, Kyomugisha A, Guthmann JP. Adherence to a six-dose regimen of artemether-lumefantrine for treatment of uncomplicated Plasmodium falciparum malaria in Uganda. Am J Trop Med Hyg. 2004 Nov;71(5):525-30. PMID 15569777
- [Background] de Vries PJ, Bich NN, Van Thien H, Hung LN, Anh TK, Kager PA, Heisterkamp SH. Combinations of artemisinin and quinine for uncomplicated falciparum malaria: efficacy and pharmacodynamics. Antimicrob Agents Chemother. 2000 May;44(5):1302-8. doi: 10.1128/AAC.44.5.1302-1308.2000. PMID 10770766
- [Derived] Achan J, Tibenderana JK, Kyabayinze D, Wabwire Mangen F, Kamya MR, Dorsey G, D'Alessandro U, Rosenthal PJ, Talisuna AO. Effectiveness of quinine versus artemether-lumefantrine for treating uncomplicated falciparum malaria in Ugandan children: randomised trial. BMJ. 2009 Jul 21;339:b2763. doi: 10.1136/bmj.b2763. PMID 19622553